CLINICAL TRIAL: NCT04861103
Title: Anticoagulation Profile in Pregnant Women Treated With Three Times a Day of Low Molecular Weight Heparin (LMWH)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Afshan B. Hameed, M.D., Maternal Fetal Medicine Physician, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20195544
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy, High Risk; Anticoagulants
MeSH Terms: interventions — Enoxaparin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Factor Xa levels in pregnant women with therapeutic Lovenox divided into three times a day dosing (Experimental): Therapeutic Lovenox dosing split into three times a day dosing for 5 day. Xa levels a measured.
  Interventions: Drug: Lovenox

INTERVENTIONS:
Drug: Lovenox — Three times a day dosing and measuring Xa peak and trough levels

SUMMARY:
Pregnancy is associated with a increased risk of developing blood clots. There is nearly a 5 times greater risk of developing a blood clot in pregnancy. Lovenox is a medication that helps to prevent the body from developing clots. It is safe to use in pregnancy. Previous studies have demonstrated that despite recommendation of Lovenox, to prevent blood clots, the majority of patient's (70 to 90%) did not receive adequate levels of Lovenox at times throughout the day, which likely increases the risk of developing clots. The increase in blood volume and increase in kidney function that occurs in pregnancy may contribute to the inadequate levels. Currently the recommendation for pregnant and nonpregnant patients requiring Lovenox, is to calculate the daily dose of Lovenox and split the dose, giving half in the morning and the other half in the evening. This research study proposes that due to changes in the body during pregnancy that the daily Lovenox dosing be split into three times a day to achieve more consistent levels of Lovenox than twice a day in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous or multiparous women with single intrauterine pregnancies who require therapeutic low molecular weight heparin during their pregnancy.
* Participants must be age 18 or older.

Exclusion Criteria:

* Women with multiples.
* Women less than age 18
* History of Heparin Induced Thrombocytopenia (HIT)
* Allergy to enoxaparin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Factor Xa levels | 4 hours after injection

CONTACTS AND LOCATIONS:
Overall Officials: Afshan Hameed, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Undecided